CLINICAL TRIAL: NCT01447420
Title: A Clinical Trial Comparing the Sustained Virological Response in Terms of Expression Profile of IL- 28B in Genotype 1 HCV-Infected Treatment-Naïve Subjects With Chronic Hepatitis C on Pegasys® (Peginterferon Alfa-2A) Plus Copegus® (Ribavirin)
Brief Title: A Study of Sustained Virological Response in Relation to IL28-b Expression in Treatment-Naïve Patients With Chronic Hepatitis C Genotype 1 on Combination Treatment With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25592
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- Peginterferon Alfa-2a Plus Ribavirin (Experimental)
  Interventions: Drug: peginterferon alfa-2a; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a — 180 mcg sc weekly, 48 weeks
Drug: ribavirin [Copegus] — 1'000 or 1'200 mg orally daily, 48 weeks

SUMMARY:
This multi-center, open-label study will evaluate the efficacy and safety of Pegasys (peginterferon alfa-2a) and Copegus (ribavirin) in relation to IL28-b gene expression in treatment-naïve patients with chronic hepatitis C genotype 1. Patients will receive Pegasys (180 mcg sc weekly) and Copegus ( 1'000 or 1'200 mg orally daily) for 48 weeks. Anticipated time of study treatment is 48 weeks, follow-up is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 and <70 years of age at initiation of treatment
* Body weight between 50 kg and 125 kg at baseline
* Chronic hepatitis C, genotype 1
* Chronic liver disease consistent with HCV infection
* Compensated liver disease (Child-Pugh Grade A)

Exclusion Criteria:

* Pregnant or lactating women, and male partners of pregnant women
* Chronic hepatitis C, genotype 2, 3, 4, 5 or 6
* Previous treatment with interferon or ribavirin
* Positive for hepatitis A, hepatitis B or HIV infection
* History or evidence of a medical condition associated with liver disease other than chronic hepatitis C
* Decompensated liver disease and/or liver disease Child-Pugh classification >6
* Hepatocellular carcinoma
* History or evidence of esophageal bleeding
* Hemoglobinopathy, or any other cause for possible hemolysis
* Hb <11 g/dL in women, <12 g/L in males

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Brazil (11):
  - Vitória, Espírito Santo
  - Salvador, Estado de Bahia
  - Juiz de Fora, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Joinville, Santa Catarina
  - Sao Jose Do Rio Preto, Santa Catarina
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Santos, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 participants were enrolled from February 2011 to November 2012 at 14 study sites in Brazil.
Groups:
- Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC: Eligible participants with interleukin 28B (IL28-B) - RS12979860 Genotype - CC, were administered peginterferon alfa-2a, 180 micrograms (mcg) subcutaneous (SC) per week plus ribavirin orally at a dose based on the initial weight (1,000 mg per day for less than (<) 75 kg and 1,200 mg per day for greater than or equal to [>=] 75 kg).
- Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT: Eligible participants with interleukin 28B (IL28-B) - RS12979860 Genotype - CT, were administered peginterferon alfa-2a, 180 mcg SC per week plus ribavirin orally at a dose based on the initial weight (1,000 mg per day for < 75 kg and 1,200 mg per day for >= 75 kg).
- Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT: Eligible participants with interleukin 28B (IL28-B) - RS12979860 Genotype - TT, were administered peginterferon alfa-2a, 180 mcg SC per week plus ribavirin orally at a dose based on the initial weight (1,000 mg per day for < 75 kg and 1,200 mg per day for >= 75 kg).
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT
Started | 39 | 72 | 18
Completed | 29 | 45 | 8
Not Completed | 10 | 27 | 10
Not completed — Adverse Event | 2 | 4 | 2
Not completed — Protocol Violation | 3 | 3 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0
Not completed — Lack of Efficacy | 1 | 19 | 8

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of any study medication.
Groups:
- Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT: Eligible participants with interleukin 28B (IL28-B) - RS12979860 Genotype - CT, were administered with peginterferon alfa-2a, 180 mcg SC per week plus ribavirin orally at a dose based on the initial weight (1,000 mg per day for < 75 kg and 1,200 mg per day for >= 75 kg).
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT | Total
Number analyzed (Participants) | 39 | 72 | 18 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.51 (12.71) | 50.43 (10.92) | 52.33 (10.22) | 50.12 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 33 | 9 | 64
  Male | 17 | 39 | 9 | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response Rate in Relation to Interleukin 28B Expression
Description: Participants with sustained virological response (SVR) rate in relation to interleukin 28B expression were reported. SVR rate is defined as the percentage of participants with undetectable HCV Ribonucleic acid (RNA), measured at least 24 weeks after the end of treatment (48 weeks) in terms of the expression profile of Interleukin 28B (IL-28B) (CC, CT or TT) in participants with genotype 1 hepatitis C virus (HCV) chronic infection. Participants with detectable HCV RNA or without measurement at the end of the follow-up period were considered as non-responders.
Time Frame: At Week 72
Population: The efficacy population included all enrolled participants who received at least one dose of any study medication, excluding one participant who took medication and had HCV RNA undetectable at Baseline (Week 0).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT
Number analyzed (Participants) | 38 | 72 | 18
Percentage of participants | 63.2 [46.0 to 78.2] | 26.4 [16.7 to 38.1] | 33.3 [13.3 to 59.0]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT; IL28B Genotypes (CC, CT or TT); Test type: Superiority or Other; p = 0.0007, Chi-squared; Participants without measurement at the end of the 24 week untreated follow-up period were considered as non-responders

2. Primary Outcome: Percentage of Participants With Incidence of Anemia
Description: Anemia is a condition marked by a deficiency of red blood cells (RBCs) or of hemoglobin (Hb) in the blood, resulting in pallor and weariness anemia (Hb < 11 gram per decilitre (g/dL) for women and Hb < 12 g/dL for men). Incidence of anemia was calculated by dividing the number of participants who experienced the event by the number of participants in the safety population.
Time Frame: Up to Week 72
Population: Safety population included all enrolled participants who received at least one dose of any study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Peginterferon Alfa-2a Plus Ribavirin: Eligible participants were administered peginterferon alfa-2a 180 mcg SC weekly, 48 weeks and Ribavirin 1,000 mg per day for < 75 kg and 1,200 mg per day for >= 75 kg, orally daily, 48 weeks
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin
Number analyzed (Participants) | 129
Percentage of participants | 67.4 [58.6 to 75.4]

3. Secondary Outcome: Number of Participants With Viral Response Rate (Rapid/Early/End of Treatment) in Relation to IL28-B Expression
Description: Viral Response rate (rapid/early/end of treatment) in relation to IL28-B expression (measured by the rate of non-detection of HCV RNA at treatment Weeks 4, 12, 24 and after the End of Treatment (EOT, i.e. Week 48) based on the expression profile of IL-28B (CC, CT or TT) were reported. Rapid virologic response (RVR) was defined as undetectable HCV RNA at treatment Week 4. Partial early virological response (pEVR) was defined as positive HCV viral load, but with a >= 2 log10 international units (IU) per millilitre (mL) reduction at treatment Week 12 from Baseline (Week 0); Complete early virologic response (cEVR) was defined as undetectable HCV RNA at treatment Week 12; Virologic response at treatment Week 24 (VR 24) was defined as undetectable HCV RNA at treatment Week 24; Virologic response at end of treatment (EOT) was defined as undetectable HCV RNA at treatment Week 48; SVR at 24 weeks after end of treatment was defined as undetectable HCV RNA at 24 weeks after EOT.
Time Frame: Weeks 4, 12, 24, 48, 60 and 72
Population: The efficacy population included all enrolled participants who received at least one dose of any study medication, excluding one participant who took medication and had HCV RNA undetectable at baseline.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT
Number analyzed (Participants) | 38 | 72 | 18
participants
  RVR rate, Week 4 (n = 14) | 11 | 3 | 0
  pEVR rate, Week 12 (n = 33) | 4 | 24 | 5
  cEVR rate, Week 12 (n = 72) | 31 | 36 | 5
  VR rate, Week 24 (n = 87) | 31 | 46 | 10
  VR rate, EOT (Week 48) (n = 74) | 28 | 37 | 9
  VR rate, 12 weeks post-treatment (n = 50) | 25 | 19 | 6
  SVR rate, 24 weeks or more post-treatment (n = 49) | 24 | 19 | 6

4. Secondary Outcome: Number of Participants With Sustained Virological Response and Occurrence of Anemia During The First Month of Treatment and After the First Month of Treatment
Description: Participants with sustained virological response (SVR) and development of anemia during the first month and after the first month of treatment according to the different expression profiles of IL-28B were reported.
Time Frame: Up to Week 72
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT
Number analyzed (Participants) | 38 | 72 | 18
participants
  SVR with No anemia (n = 15, 20, 6) | 9 | 4 | 2
  In the first month of treatment (n = 10, 15, 2) | 6 | 3 | 0
  After the first month of treatment (n = 13, 37,10) | 9 | 12 | 4
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT; Anemia after the first month of treatment vs No anemia; Test type: Superiority or Other; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.69 to 4.14] — Odds Ratio for SVR estimated from the logistic regression model
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT; Anemia in the first month of treatment vs No anemia; Test type: Superiority or Other; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.28 to 2.59] — Odds Ratio for SVR estimated from the logistic regression model
Statistical Analysis 3: Comparison: Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT; IL28B - CC vs CT; Test type: Superiority or Other; Odds Ratio (OR) = 5.45, 95% CI 2-sided [2.27 to 13.12] — Odds Ratio for SVR estimated from the logistic regression model
Statistical Analysis 4: Comparison: Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC vs Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT; IL28B - CC vs TT; Test type: Superiority or Other; Odds Ratio (OR) = 4.03, 95% CI 2-sided [1.19 to 13.61] — Odds Ratio for SVR estimated from the logistic regression model

5. Secondary Outcome: Number of Participants With Viral Load Reduction (HCV-RNA Levels) at Week 4 and 12
Description: Viral load reduction at Week 4 and Week 12 relative to the Baseline (Week 0) in terms of the expression profile of IL-28b was reported. The reduction was measured according to the following ranges: < 1.0 log IU/ml; >= 1.0 and < 2.0 log IU/ml; >= 2.0 and < 3.0 log IU/ml; >= 3.0 and <4.0 log IU/ml; >= 4.0 log IU/ml. Changes in viral load are usually reported as a log change (in powers of 10). For example, a two log decrease in viral load (2 Log10) is a decrease of 10^2 or 100 times to the previously reported levels. N = number of participants, for Week 0 to Week 4 (n = 34, 68, 17) and Week 0 to Week 12 (n = 35, 69, 18) for CC, CT and TT genotypes respectively.
Time Frame: From Baseline (Week 0) to Week 12
Population: The efficacy population included all enrolled participants who received at least one dose of any study medication, excluding one participant who took medication and had HCV RNA undetectable at baseline. Participants with available data at the time of evaluation were analyzed.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CC | Peginterferon Alfa-2a Plus Ribavirin With Genotype - CT | Peginterferon Alfa-2a Plus Ribavirin With Genotype - TT
Number analyzed (Participants) | 35 | 69 | 18
participants
  Week 0 - Week 4 (<1.0 log10 UI / ml) | 0 | 26 | 10
  Week 0 - Week 4 (>=1.0 e < 2.0 log10 UI / ml) | 4 | 24 | 5
  Week 0 - Week 4 (>=2.0 e < 3.0 log10 UI / ml) | 9 | 13 | 1
  Week 0 - Week 4 (>=3.0 e < 4.0 log10 UI / ml) | 13 | 2 | 1
  Week 0 - Week 4 (>=4.0 log10 UI / ml) | 8 | 3 | 0
  Week 0 - Week 12 (<1.0 log10 UI / ml) | 0 | 1 | 3
  Week 0 - Week 12 (>=1.0 e < 2.0 log10 UI / ml) | 3 | 9 | 5
  Week 0 - Week 12 (>=2.0 e < 3.0 log10 UI / ml) | 5 | 11 | 3
  Week 0 - Week 12 (>=3.0 e < 4.0 log10 UI / ml) | 5 | 22 | 3
  Week 0 - Week 12 (>=4.0 log10 UI / ml) | 22 | 26 | 4

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: Adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant that administers a pharmaceutical product, which does not necessarily have a causal relationship with treatment. Safety population was used which included all enrolled participants who received at least one dose of any study medication.
Groups:
- Peginterferon Alfa-2a Plus Ribavirin: Eligible participants were administered peginterferon alfa-2a, 180 mcg SC weekly, 48 weeks and Ribavirin 1000 mg per day for < 75 kg and 1200 mg per day for >= 75 kg, orally daily, 48 weeks.
Arm/Group | Peginterferon Alfa-2a Plus Ribavirin
Serious Adverse Events (participants affected / at risk) | 6/129
Other Adverse Events (participants affected / at risk) | 125/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a Plus Ribavirin (N=129)
Chest pain (Cardiac disorders) | 1
Optic ischaemic neuropathy (Eye disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Perianal erythema (Gastrointestinal disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a Plus Ribavirin (N=129)
Anaemia (Blood and lymphatic system disorders) | 41
Neutropenia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Dizziness (Cardiac disorders) | 15
Eye pain (Eye disorders) | 9
Nausea (Gastrointestinal disorders) | 32
Diarrhoea (Gastrointestinal disorders) | 25
Dyspepsia (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 15
Upper abdominal pain (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Aphthous stomatitis (Gastrointestinal disorders) | 8
Pyrexia (General disorders) | 48 — General disorders and administration site conditions
Asthenia (General disorders) | 35 — General disorders and administration site conditions
Fatigue (General disorders) | 20 — General disorders and administration site conditions
Discomfort (General disorders) | 17 — General disorders and administration site conditions
Pain (General disorders) | 15 — General disorders and administration site conditions
Influenza (Infections and infestations) | 54
Decreased appetite (Metabolism and nutrition disorders) | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 42
Chills (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 55
Insomnia (Psychiatric disorders) | 25
Irritability (Psychiatric disorders) | 25
Depression (Psychiatric disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 25
Alopecia (Skin and subcutaneous tissue disorders) | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8
Epistaxis (Vascular disorders) | 7
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.